CLINICAL TRIAL: NCT00487201
Title: Endoscopic Treatment of Biliary Strictures After LTX: Balloon Dilatation Versus Stent Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120-2006
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2007-06-18 (Estimated); Status verified 2007-05

CONDITIONS: Biliary Obstruction; Biliary Stenosis; Biliary Stricture
Keywords: liver transplantation; biliary strictures; ERCP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: endoscopic balloon dilatation
Procedure: plastic stent placement

SUMMARY:
Background and Study Aims: Biliary strictures are a major cause of morbidity following liver transplantation with an overall incidence between 10 and 30 %. Up to now biliary strictures were dilated subsequently one to three plastic stents with a diameter of eight to ten F were inserted. In general, stents were exchanged in two to three months intervals over one year. In the present prospective controlled study, efficacy and complication rates of balloon dilation have been compared with dilation plus stenting.

Patients and Methods: XY patients with high-grade biliary strictures (anastomotic and non-anastomotic) were enrolled in this prospective study in random order. X patients were treated by endoscopic balloon dilatation and Y by balloon dilatation plus plastic stent placement in six to eight weeks intervals. The primary end point was permanent opening of the biliary obstruction of 12 months. Number of endoscopic interventions and complications of the procedures were monitored.

DETAILED DESCRIPTION:
Endoscopic treatment was performed by experienced endoscopists who had each performed more than 1000 ERCP procedures. The procedure was performed with the patient under general anesthesia with propofol. A stenosis was considered to be present if the cholangiogram showed strictures with a narrowing of the anastomosis or the proximal donor duct site of the anastomosis and incomplete distal runoff of the contrast agent.

The patients were divided into two groups: 1) balloon dilatation of the stricture, 2) balloon dilatation plus plastic stent placement.

In both groups, endoscopic treatment of the patients comprised sphincterotomy, consecutive dilation of stenosis up to 10 F, removement of occluding material from choledochus duct using a balloon catheter if necessary, and repetitive balloon dilatation of the anastomosis stricture or of the non-anastomotic proximal donor duct stricture to 18 F at the first intervention and to 24 F in the following interventions.

The second group of the patients were additionally treated by large-diameter (10 F) plastic stent placement after balloon dilatation. This procedure was repeated in 6 - 8 weeks intervals in both groups.

ELIGIBILITY:
Inclusion Criteria:

* liver transplanted patients with diagnosis of biliary obstruction based on endoscopic cholangiopancreaticography older than 18 years male and female

Exclusion Criteria:

* patients with multiple organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-04; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Permanent opening of the biliary obstruction. | 12 months

SECONDARY OUTCOMES:
number of endoscopic interventions and complications of the procedures | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Kulaksiz, PD Dr., Principal Investigator — Medizinische Universitätsklinik Ulm, Innere Medizin I
Locations (2):
- Germany (2):
  - Uniklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Medizinische Universitätsklinik Ulm, Ulm, Baden-Wurttemberg

REFERENCES:
- [Background] Graziadei IW, Wiesner RH, Batts KP, Marotta PJ, LaRusso NF, Porayko MK, Hay JE, Gores GJ, Charlton MR, Ludwig J, Poterucha JJ, Steers JL, Krom RA. Recurrence of primary sclerosing cholangitis following liver transplantation. Hepatology. 1999 Apr;29(4):1050-6. doi: 10.1002/hep.510290427. PMID 10094945
- [Background] Sossenheimer M, Slivka A, Carr-Locke D. Management of extrahepatic biliary disease after orthotopic liver transplantation: review of the literature and results of a multicenter survey. Endoscopy. 1996 Sep;28(7):565-71. doi: 10.1055/s-2007-1005556. No abstract available. PMID 8911805